CLINICAL TRIAL: NCT06390618
Title: Investigation of the Biopsychosocial Effectiveness of Different Exercise Trainings in Earthquake Survivors With Post-Traumatic Stress Disorder
Brief Title: Biopsychosocial Effectiveness of Exercise Trainings in Earthquake Survivors With Post-Traumatic Stress Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erkin Oğuz SARI (Other)
Responsible Party: Sponsor-Investigator, Erkin Oğuz SARI, Research Assistant, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HKU-FTR-EOS-01
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-Traumatic Stress Disorder; Aerobic Exercise; Biopsychosocial Models; Qualitative and Quantitative Evaluation; Physical therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Exercise; Population Groups

STUDY DESIGN:
Intervention Model Description: According to randomization, they will be divided into 3 groups: aerobic exercise group (AE), combined exercise (CE) group in which biopsychosocial exercise is performed in addition to aerobic exercise, and control group (C).
Who Masked: Investigator, Outcomes Assessor
Masking Description: After the data are collected, a randomized controlled double-blind study will be conducted by ensuring the blindness of the evaluator and the statistician. Blinding will be achieved by assigning numbers to randomized patients and keeping the evaluator and statistician from knowing which patient is in which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Group (AE) (Active Comparator): A moderate intensity (50-60%) aerobic exercise program will be applied 3 days a week, using the karvonen method for aerobic exercise. According to the aerobic exercise intensity karvonen method, the formula "(Maximal Heart Rate (220-years) - Resting Heart Rate) x 50-60% + Resting Heart Rate)" will be used. 1-4. week 50%, 5-8. Exercise intensity will be increased by 60% per week.
  Interventions: Other: Aerobic Exercise (AE) Group
- Combined Exercise (CE) Group (Active Comparator): The group in which biopsychosocial exercise is performed in addition to aerobic exercise is the combined exercise (CE) group. Cognitive Exercise Therapy Approach (BETY) will be applied with group exercise as a biopsychosocial exercise. In the BETY biopsychosocial model, it is aimed to achieve biological recovery with function-oriented trunk stabilization exercises, psychological recovery by expressing negative-positive thoughts during the exercises and emphasizing staying in positive thoughts, and social recovery through group treatment.
  Interventions: Other: Combined Exercise (CE) Group
- Control Group (C) (No Intervention): There will be no intervention in the control group. The change over time in the control group and individuals with post-traumatic stress disorder will be monitored.

INTERVENTIONS:
Other: Aerobic Exercise (AE) Group — A total of 24 sessions of aerobic exercise will be performed in 8 weeks, 3 days a week.
  For aerobic exercise, a moderate intensity (50-60%) aerobic exercise program will be applied using the karvonen method. According to the aerobic exercise intensity karvonen method, the formula "(Maximal Heart Rate (220-years) - Resting Heart Rate) x 50-60% + Resting Heart Rate)" will be used. 1-4. week 50%, 5-8. Exercise intensity will be increased by 60% per week.
  Arms: Aerobic Exercise Group (AE)
Other: Combined Exercise (CE) Group — In the combined exercise group, biopsychosocial exercise will be performed in addition to aerobic exercise.
  In the combined exercise group, in addition to aerobic exercise (3, 8 weeks, 24 sessions of aerobic exercise per week), 16 sessions of biopsychosocial-based group exercise treatment will be performed 2 days a week for a total of 8 weeks.
  BETY approach will be used in group exercise treatment.
  Other Names: Cognitive Exercise Therapy Approach (BETY)
  Arms: Combined Exercise (CE) Group

SUMMARY:
In study, the investigators aim to demonstrate the effectiveness of biopsychosocial-based exercise approach in post-traumatic stress disorder of physiotherapists in post-earthquake disaster management.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of aerobic exercise and biopsychosocial exercise in addition to aerobic exercise on functional capacity, trauma symptoms, depression, anxiety, stress, sleep quality, quality of life and biopsychosocial status in earthquake victims with post-traumatic stress disorder (PTSD).

Individuals will be randomized using the covariate adaptive randomization method. According to this randomization, they will be divided into 3 groups: aerobic exercise group (AE), combined exercise (CE) group, in which biopsychosocial exercise is performed in addition to aerobic exercise, and control group (C).

A total of 16 sessions of treatment will be performed in 8 weeks, 2 days a week. In the control group, no intervention will be made. The change over time in the control group and individuals with post-traumatic stress disorder will be monitored.

Questionnaires for quantitative data before treatment and 8 weeks after treatment; Data will also be collected through interview questions for qualitative data about experience/change after 8 weeks of treatment. In our study, mixed methods research will be used because it is thought that the survey data can be more descriptive and meaningful by supporting qualitative interview questions. Explanatory sequential mixed methods type will be used as a mixed methods research design. According to this design, quantitative data will be collected first and then qualitative data about the topic to be focused on will be collected from group interviews with semi-structured interview questions. Phenomenology research focuses on the experiences of participants. Phenomenological research method will be used in qualitative research.

A moderate intensity (50-60%) aerobic exercise program will be applied 3 days a week, using the karvonen method for aerobic exercise. According to the aerobic exercise intensity karvonen method, the formula "(Maximal Heart Rate (220-years) - Resting Heart Rate) x 50-60% + Resting Heart Rate)" will be used. 1-4. week 50%, 5-8. Exercise intensity will be increased by 60% per week.

Cognitive Exercise Therapy Approach (BETY) will be applied as a biopsychosocial exercise. BETY method is a patient-centered biopsychosocial approach and a holistic treatment option. On the basis of the BETY session, warm-up movements, exercises and cooling movements will be performed sequentially. While authentic movements are performed accompanied by music as dance therapy during the warm-up and cool-down period, functional trunk stabilization exercises are used during the exercises period. In addition, cognitive change is aimed by expressing positive and negative emotions during side lying exercises. Social support will also be provided by holding BETY sessions as a group. Thus, the aim is biological recovery with exercises, psychological recovery by expressing negative-positive thoughts during exercises and emphasizing staying in positive thoughts, and social recovery with group treatment.

After the data are collected, a randomized controlled double-blind study will be conducted by ensuring the blindness of the evaluator and the statistician. Blinding will be achieved by assigning numbers to randomized patients and keeping the evaluator and statistician from knowing which patient is in which group. To calculate the sample size, power analysis will be made by referring to similar studies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with earthquake-related post-traumatic stress disorder (PTSD)
* 18-65 years old
* Individuals who agree to participate in the study voluntarily

Exclusion Criteria:

* Individuals with another psychiatric diagnosis
* Individuals with a body mass index of more than 35 kg/m2
* Individuals with a history of another trauma
* Pregnant women
* Individuals with neurological findings
* Individuals with malignancy, rheumatological, metabolic bone disease
* Individuals with a history of columna vertebralis and lower extremity surgery
* Individuals with severe osteoporosis
* Individuals who are illiterate and have communication problems
* Individuals with hearing problems
* Individuals who do not attend treatment regularly
* Individuals continuing another physiotherapy program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire (BETY-BQ) | eight weeks
  BETY-BQ scale consists of 30 different items. The five-point Likert system of the BETY scale evaluates dimensions such as pain, functionality, mood, sociability, sexuality and sleep quality. Each of the items in the scale is scored between 0-4. The survey is scored between 0-120, and a higher score indicates a poor biopsychosocial situation.
Qualitative Interview Questions (from group interviews with semi-structured interview questions) | eight weeks
  In group interviews, semi-structured interview questions will be asked and voice recordings will be made. Afterwards, the voice recordings will be analyzed.

SECONDARY OUTCOMES:
6 Minute Walking Test | eight weeks
  Functional capacity is evaluated with the 6 Minute Walk Test (6MWT). The test is applied in a 30 m corridor. Before starting the test, patients are asked to walk as fast as they can without running, and are told that they can rest if they feel too short of breath and/or tired, and that the time they rest is included in the test. Before, after and at the first minute of the test, patients' blood pressure, heart rate and oxygen saturation are evaluated with pulse oximetry, and their perceptions of shortness of breath, fatigue and leg fatigue are evaluated with the Modified Borg Scale.
  The total distance the patient was able to walk after the test was recorded and will be expressed as a percentage of what was expected.
Post-Traumatic Stress Disorder (PTSD) Checklist (PCL-5) | eight weeks
  The PCL-5 is an easily administered self-report measure that maps 20 symptoms of PTSD outlined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). The 20-item self-report measure of PTSD, which is rated on a five-point scale (scored 0-4) and yields a scale score range of 0-80, was expanded from the previous PCL.
  The PCL-5 consists of four scales that map PTSD symptom clusters in the DSM-5: reexperiencing (criteria B), avoidance (criteria C), negative changes (criteria D), and hyperarousal (criteria E).
  Although the cut-off score of 47 seems appropriate for clinical use, it is thought that using a score of 48 is more reliable in distinguishing individuals with PTSD in community samples.
  With the adaptation made by Weathers et al., the items of the scale were increased to 20 items, compatible with PTSD symptoms (Waethers 2013). The adaptation study of PCL in Turkey was carried out by Boysan and his colleagues (Boysan 2017).
Post-Traumatic Stress Diagnostic Scale (PTSDS) | eight weeks
  The scale developed to determine post-traumatic stress disorder is a self-report scale consisting of fifty items. The scale was developed by Foa et al. It is possible to identify people who meet the diagnosis of PTSD and measure the severity of symptoms with the help of a scale with structure and content prepared according to DSM-IV diagnostic criteria. The scale was adapted into Turkish by Işıklı. A total score of 1-10 is considered mild symptoms, 11-20 is considered moderate symptoms, 21-35 is considered moderate-severe symptoms, and scores of 36 and above are considered severe symptoms.
Impact of Events Scale-Revised (IES-R) | eight weeks
  The Impact of Events Scale-R was used to measure post-traumatic symptom severity. The scale was developed by Horowitz et al. to assess subjective distress caused by traumatic events. Depending on the changes in the clinical situation over time, new items from Weiss and Marmar were added to the scale, and the new scale, which increased to 21 items and had three sub-factors, was named Event Impact Scale-R. These sub-dimensions; re-experiencing, avoidance and hyperarousal. It is a self-report scale that measures post-traumatic stress level, adapted into Turkish by Çorapçıoğlu et al.
  A scale score of up to 24 points is considered normal, 24 and above is considered partial PTSD, 33 and above is considered the best limit for possible PTSD, and 37 and above is considered PTSD high enough to suppress the immune system.
Depression Anxiety and Stress Scale (DASS-21) | eight weeks
  DASS-21 is the short form of the Depression, Stress and Anxiety Scale, developed by Lovibond and Lovibond, consisting of 42 items. The Turkish reliability and validity study of the scale was conducted by Yılmaz, Boz and Arslan in 2017.
  DASS-21 has three subscales: depression, stress and anxiety; There are seven questions in each dimension. The scale is a 4-point Likert type scale (0-Not suitable for me, 1-Sometimes suitable for me, 2-Usually suitable for me and 3-Completely suitable for me). The scores that can be obtained from each subscale vary between 0 and 21. A high score means that you have high levels of depression/anxiety/stress symptoms. If an individual scores 5 points or more on the depression subscale, 4 points or more on the anxiety subscale, and 8 points or more on the stress subscale, it indicates that he or she has a relevant problem.
Pittsburgh Sleep Quality Index (PSQI) | eight weeks
  The Pittsburgh Sleep Quality Index (PSQI) was developed by Buysse and his team. It was adapted into Turkish by Ağargün et al. in 1996. PSQI is a feedback scale that evaluates sleep quality and disorder over the past month and consists of 24 questions in total.
  Seven sub-dimensions, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorder, use of sleeping pills, and daytime dysfunction, are evaluated with 19 questions answered by the adult individual. The sum of the scores on the seven subscales gives the total PSQI score. The score of each subscale varies between 0 and 3. The total PSQI score varies between 0-21. Sleep quality of those with a total score of 5 or less is considered good.
SF-36 Short Form | eight weeks
  The survey contains 36 items. The survey measures health-related quality of life under eight subheadings. It gives results for 8 parameters consisting of physical function, physical role difficulty, emotional role difficulty, energy-vitality-vitality, mental health, social functionality, pain and general health perception. It also allows comparison of current health status with last year in the last item it contains. The scores from each subheading are summed to obtain a score between 0 (poor quality of life) and 100 (good quality of life).
  The Turkish validity of the scale used was conducted by Koçyiğit et al. in 1999.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adhikari SP, Bimali I, Baidya S, Shakya NR. Community-based rehabilitation for physically impaired earthquake victims: An evidence-based practice protocol and its pre-post experimental study. J Family Med Prim Care. 2018 Nov-Dec;7(6):1327-1333. doi: 10.4103/jfmpc.jfmpc_112_18. PMID 30613520
- [Result] Ahmed SK, Dhama K, Abdulqadir SO, Omar RM, Ahmed DR, Chakraborty C, Saied AA. The mental health of people in Turkey-Syria earthquake-affected areas needs urgent attention. Asian J Psychiatr. 2023 Jun;84:103573. doi: 10.1016/j.ajp.2023.103573. Epub 2023 Mar 28. No abstract available. PMID 37028233
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Gibbons WJ, Fruchter N, Sloan S, Levy RD. Reference values for a multiple repetition 6-minute walk test in healthy adults older than 20 years. J Cardiopulm Rehabil. 2001 Mar-Apr;21(2):87-93. doi: 10.1097/00008483-200103000-00005. PMID 11314289
- [Result] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Result] Kukihara H, Yamawaki N, Uchiyama K, Arai S, Horikawa E. Trauma, depression, and resilience of earthquake/tsunami/nuclear disaster survivors of Hirono, Fukushima, Japan. Psychiatry Clin Neurosci. 2014 Jul;68(7):524-33. doi: 10.1111/pcn.12159. Epub 2014 Mar 4. PMID 24444298
- [Result] Kuroda Y, Iwasa H, Orui M, Moriyama N, Suemoto CK, Yashiro C, Matsuda K, Yasumura S. Risk Factor for Incident Functional Disability and the Effect of a Preventive Exercise Program: A 4-Year Prospective Cohort Study of Older Survivors from the Great East Japan Earthquake and Nuclear Disaster. Int J Environ Res Public Health. 2018 Jul 6;15(7):1430. doi: 10.3390/ijerph15071430. PMID 29986471
- [Result] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Result] Manger TA, Motta RW. The impact of an exercise program on posttraumatic stress disorder, anxiety, and depression. Int J Emerg Ment Health. 2005 Winter;7(1):49-57. PMID 15869081
- [Result] Momma H, Niu K, Kobayashi Y, Huang C, Otomo A, Chujo M, Tadaura H, Nagatomi R. Leg extension power is a pre-disaster modifiable risk factor for post-traumatic stress disorder among survivors of the Great East Japan Earthquake: a retrospective cohort study. PLoS One. 2014 Apr 23;9(4):e96131. doi: 10.1371/journal.pone.0096131. eCollection 2014. PMID 24760054
- [Result] Thordardottir K, Gudmundsdottir R, Zoega H, Valdimarsdottir UA, Gudmundsdottir B. Effects of yoga practice on stress-related symptoms in the aftermath of an earthquake: A community-based controlled trial. Complement Ther Med. 2014 Apr;22(2):226-34. doi: 10.1016/j.ctim.2014.01.008. Epub 2014 Feb 2. PMID 24731893
- [Result] Tian Y, Wong TK, Li J, Jiang X. Posttraumatic stress disorder and its risk factors among adolescent survivors three years after an 8.0 magnitude earthquake in China. BMC Public Health. 2014 Oct 15;14:1073. doi: 10.1186/1471-2458-14-1073. PMID 25318533
- [Result] Tsuji T, Sasaki Y, Matsuyama Y, Sato Y, Aida J, Kondo K, Kawachi I. Reducing depressive symptoms after the Great East Japan Earthquake in older survivors through group exercise participation and regular walking: a prospective observational study. BMJ Open. 2017 Mar 3;7(3):e013706. doi: 10.1136/bmjopen-2016-013706. PMID 28258173
- [Result] Zahid M, Unal E, Ozdemir Isik O, Oksuz S, Karakaya J, Erguney Cefle A. The reliability, validity, and responsiveness of Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire for patients with fibromyalgia. Int J Rheum Dis. 2022 Jun;25(6):685-691. doi: 10.1111/1756-185X.14325. Epub 2022 May 3. PMID 35505570